CLINICAL TRIAL: NCT01592903
Title: Identification and Characterization of Putative Leiomyoma Stem Cells.
Brief Title: Somatic Stem Cells in Leiomyomas?
Status: Completed | Type: Observational
Sponsor: Igenomix (Industry)
Responsible Party: Principal Investigator, Carlos Simon, Director of Clinical Research IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Other Study IDs: 1006-C-072-CS-F
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Leiomyomas
Keywords: Uterine fibroids; somatic stem cell; Side Population
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PHASE 1:SAMPLE COLLECTION Duration: From the first month to 36th month approximately. PHASE 2: CELL PREPARATION PROTOCOL Duration: From the first month to 12th month PHASE 3: ISOLATION OF PUTATIVE SOMATIC STEM CELLS Duration: From the third month (March 2010) to 12th month PHASE 4: CELL CULTURE Duration: From the sixth month to 18th month PHASE 5: ENDOCRINE CHARACTERIZATION Duration:From the 18th month to 36th month Biospecimen Retention Samples With DNA - samples retained, with potential for extraction of DNA from at least one of the types of samples retained (e.g., frozen tissue, whole blood) Biospecimen Description Samples of human leiomyomas obtained from patients with symptomatic uterine fibroids.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with symptomatic uterine fibroids.: Samples of human leiomyomas are obtained from patients undergoing laparoscopic myomectomy for symptomatic uterine fibroids. These leiomyomas are isolated and cultured for stem cells.
  Interventions: Genetic: Laparoscopic myomectomy. Following analysis and proliferation of cells isolated from removed human leiomyoma.

INTERVENTIONS:
Genetic: Laparoscopic myomectomy. Following analysis and proliferation of cells isolated from removed human leiomyoma. — * Obtention of one part of removed human leiomyoma after surgery and maintained in 4ºC until procedures.
  * Sample digestion through controlled enzymes.
  * Isolated the "Side Population" from leiomyoma cell suspension by Flow cytometry .
  * Culture of these cells.
  * Morphological and genetic characterization.
  * Assessment of pluripotent potential from isolated cells.
  * Analysis of the degree of functionality.

SUMMARY:
The purpose of this study is to identify and characterize the Somatic Stem Cell (SSC) responsible for the formation and growth of leiomyomas using the Side Population method.

DETAILED DESCRIPTION:
The organ of interest in our study is the myometrium, a muscle layer of the uterus located between the perimetry and the endometrium.

The investigators try to identify, locate and characterize the myometrial stem cell population in the uterine fibroids by isolation of "Side Population" by flow cytometry. Once the investigators achieve the purposes to set out, the investigators would try to maintain "in vitro" stem cell population isolated from myometrial fibroids, for further endocrine characterization. Finally, the investigators would try to induce the formation of fibroids in murine models as a first step to demonstrate that the origin of these formations is due to the abnormal proliferation of myometrial adult stem cells. The results of this study will allow the identification of the cell population in the fibroids. The investigators also can being able to compare with the myometrium in order to establish a relationship that helps us to understand more about the pathophysiology of this disease, using these stem cells as targets therapy in the treatment of this myometrium condition.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis for subserosal, intramural and submucosal fibroids.
* Aged between 20 and 40 years
* Signing of informed consent for collection and storage of biological samples.

Exclusion criteria:

* Contraindications for surgery.
* Failure to sign informed consent for collection and storage of biological samples.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female patients from 20 years and older undergoing laparoscopic myomectomy for symptomatic uterine fibroids.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Formation and growth of human leiomyomas | 36 months
  Assessment of pluripotent potential from isolated cells responsible for the formation and growth of human leiomyomas.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simon, MDPhD, Principal Investigator — Igenomix
Locations (1):
- IVI Valencia, Valencia, Valencia, Spain